CLINICAL TRIAL: NCT07387484
Title: Effect of Patient Position on Dermatomal Spread and Analgesic Outcomes of Erector Spinae Plane Block in Thoracic Surgery: A Prospective Randomized Clinical Trial
Brief Title: Effect of Patient Position on Erector Spinae Plane Block in Thoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ekin Guran, MD, Principal investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP_position
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thoracic Surgery, Video Assisted; Postoperative Pain
Keywords: video assisted thorachoscopic surgery; erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Parapsychology; Dental Occlusion; Bupivacaine; Sitting Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting Position Group (Active Comparator): Intervention: Erector Spinae Plane Block Ultrasound-guided unilateral erector spinae plane block performed in the sitting position using 30 mL of 0.25% bupivacaine.
  Interventions: Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) sitting position
- Lateral Decubitus Position Group (Experimental): Intervention: Erector Spinae Plane Block Ultrasound-guided unilateral erector spinae plane block performed in the lateral decubitus position (operative side up) using 30 mL of 0.25% bupivacaine.
  Interventions: Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) lateral position

INTERVENTIONS:
Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) sitting position — Erector spinae plane block-sitting position
  Arms: Sitting Position Group
Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) lateral position — Erector Spinae Plane Block-Lateral position
  Arms: Lateral Decubitus Position Group

SUMMARY:
The erector spinae plane (ESP) block is a widely used regional anesthesia technique for postoperative analgesia in thoracic surgery. The block can be performed in different patient positions, most commonly sitting or lateral decubitus, but the effect of patient position on dermatomal sensory spread and analgesic efficacy has not been clearly established.

This prospective, randomized, single-blind clinical trial aims to compare the effects of ESP block performed in sitting versus lateral decubitus position on dermatomal sensory distribution and postoperative analgesic outcomes in patients undergoing video-assisted thoracic surgery.

DETAILED DESCRIPTION:
Adult patients scheduled for elective video-assisted thoracic surgery will be randomly assigned to receive ultrasound-guided unilateral erector spinae plane block either in the sitting position or in the lateral decubitus position. In both groups, the block will be performed at the same thoracic level using 30 mL of 0.25% bupivacaine under ultrasound guidance.

Dermatomal sensory spread will be assessed 15 minutes after block placement using cold sensation (alcohol-soaked cotton) and pin-prick testing. Postoperative analgesia will be standardized in all patients using patient-controlled analgesia with tramadol. Pain scores and opioid consumption will be recorded during the first 24 postoperative hours.

The primary outcome is the extent of dermatomal sensory spread. Secondary outcomes include postoperative pain scores, time to first rescue analgesic, and total opioid consumption within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* ASA physical status II-IV
* Scheduled for elective video-assisted thoracic surgery
* Ability to provide written informed consent

Exclusion Criteria:

* Known allergy to local anesthetics
* Chronic opioid use
* Preexisting chronic pain
* Severe cognitive impairment
* Technical difficulty with positioning
* Emergency surgery
* Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Dermatomal sensory spread | 15 minutes after the block application
  Cranial and caudal sensory limits and total number of dermatomes affected, assessed by cold sensation and pin-prick testing.

SECONDARY OUTCOMES:
Postoperative pain scores (Numeric Rating Scale) | Postoperative 0, 2, 6, 12, and 24 hours
  Numeric Rating Scale, 0-10 points, 0=no pain, 10= worst pain imaginable
Total opioid consumption | First 24 postoperative hours

IPD SHARING:
Plan to Share IPD: Yes